CLINICAL TRIAL: NCT02572440
Title: Department of Anesthesiology, Beijing Anzhen Hospital, Capital Medical University
Brief Title: Autologous Platelet-rich Plasma (aPRP) for Complex Aortic Arch Surgerymacrovascular Operation
Status: Temporarily not available | Type: Expanded Access
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Zhao Liyun, Vice-president anesthesiology department Beijing Anzhen Hospital, Beijing Anzhen Hospital
Other Study IDs: Z13110700213134
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Autologous Blood Transfusion
Keywords: Aortic arch surgery; Blood conservation; aPRP

INTERVENTIONS:
Procedure: Sorin XTRA/Sorin Group,

SUMMARY:
Perioperative blood loss continues to be a serious problem in complex aortic arch surgery using deep hypothermic circulatory arrest (DHCA). Major blood loss causes increased morbidity and mortality [1]. These patients often require transfusion of allogeneic blood products. It has been estimated shortages of blood supply in China will worsen [2]. Clinicians have made significant progress to decrease the quality of allogenic blood transfusion.

Increasing postoperative hemorrhage risk of aortic arch patients undergoing DHCA may be related to CPB induced hemostatic defect, the use of the CPB is likely to contribute to coagulation factor lost and platelet dysfunction [3, 4]. We are aware of the potential benefit of aPRP, withdrawal of aPRP immediately before initiating CPB appears to be a promising approach because it avoids CPB-related platelet damage and limits post-CPB blood loss. So we adopted and used aPRP as a blood conservation technique to reduce blood transfusion in aortic arch surgery with DHCA. Autologous red blood cells were infused to maintain a HGB level above 100 g/L after heparin neutralizing activity. And aPRPs were transfused after heparin neutralizing activity as no active bleeding was observed. Our goal was to determine the effect between aPRP and homologous transfusion on perioperative bleeding during complex aortic arch surgery using DHCA.

DETAILED DESCRIPTION:
1. Patient selection 42 type A aortic dissections patients were asked to participate in a prospective, randomized trial comparing aPRP technique with regular blood conservation. 6 patients were excluded The patients were randomized into two groups: regular blood conservation group(n=18) and aPRP group(n=18). Patients gave informed consent, and ethical permission was approved by the Human Ethics Committee of Beijing Anzhen Hospital. The grouping situation is blinded to the surgeon, perfusionist and statistician.
2. Anesthesia and monitoring method All patients were monitored according to the American Society of Anesthesia guidelines and received standard general anesthesia. A post-operative analgesic pump was used until four days after surgery. The same group of surgeons performed all operations. Extracorporeal circulation used DHCA and axillary arterial anterograde cerebral perfusion. In addition, the same group of physicians managed extracorporeal circulation.
3. Autologous Platelet-Rich Plasma Harvest Technique In the treatment group, shortly after administration of general anesthesia, blood was collected via central venous catheter 60 ml per minute (that was proven to be safe) and approximately 15-20 mL/kg of whole blood was collected. The harvested blood was then centrifuged at 2400 rpm to separate the red blood cells (RBC) from the autologous platelet rich plasma (aPRP). The separated blood component was processed by acid sodium citrate glucose solution (AcD-A) for anti-coagulation. No systemic heparin was administered at this time. The aPRP component was then stored at 20℃ - 24℃. When the blood withdrawal was proceeding, lactated ringer's solution and succinylated gelatin were used via the peripheral vein to dilate circulating capacity and maintain hemodynamic stability. A vasoactive drug was used if necessary. The systematic heparinization began after blood collection had completed. General blood salvage was performed during surgery and transfused according to the patient's actual intraoperative needs.

   The mean quantity of whole blood collected for Autologous Platelet-Rich Plasma Harvest was 1037 ± 286 mL. The control group was only subjected to general intraoperative blood conservation using red blood cell salvage and allogenic blood transfusion.
4. Transfusion Practice Autologous red blood cells were infused to maintain the HGB level above 100 g/L. While on CPB, the hemoglobin (HGB) level was maintained between 70 g/L to 90 g/L. Salvaged blood was also used following CPB. FFP, platelets, and aPRP were transfused after protamine reversed heparinization, since no active bleeding was observed. Therapeutic transfusion triggers were: INR TEG-R>11 min for FFP administration; TEG-a <63 degrees for human fibrinogen; and TEG-MA <52 mm for aphaeresis platelets

ELIGIBILITY:
Inclusion Criteria:

* adults older than 18 years old, type A aortic dissections patients undergoing frozen elephant trunk with total arch replacement (Bentall plus Sun's surgery) with DHCA.

Exclusion Criteria:

* patients with hepatitis B virus infection, coagulation disorder, anemia (HBG<11mg/dl), stopping anticoagulants less than 7 days and end-stage renal disease dependent on hemodialysis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2014-10; Primary Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China